CLINICAL TRIAL: NCT00680381
Title: Transitional Treatment of Adolescents in Family Therapy
Acronym: Transitions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: DA15762; R01DA015762 (NIH)
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Substance Abuse
Keywords: adolescent substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Following 12 weeks of Functional Family Therapy (FFT), semi-weekly therapist phone calls for eight weeks.
  Interventions: Behavioral: MTI, Minimal Transitional Intervention
- 2 (Active Comparator): Following 12 weeks of FFT, weekly one-hour group therapy for eight weeks
  Interventions: Behavioral: GTI, Group Transitional Intervention
- 3 (Active Comparator): Following 12 weeks of FFT, an eight-week, customized series of therapist visits with the adolescent, family, teachers, coaches and others who can support the adolescent's reduced level of drug use.
  Interventions: Behavioral: STI, Systems Transitions Intervention

INTERVENTIONS:
Behavioral: MTI, Minimal Transitional Intervention — Following 12 weeks of Functional Family Therapy (FFT), semi-weekly phone calls from a therapist for eight weeks.
  Arms: 1
Behavioral: GTI, Group Transitional Intervention — Following 12 weeks of FFT, weekly one-hour sessions of group therapy for eight weeks.
  Arms: 2
Behavioral: STI, Systems Transitions Intervention — Following 12 weeks of FFT, an individualized eight-week series of therapist meetings with the adolescent, family, police, teachers, coaches and others who can support the adolescent's reduced drug use.
  Arms: 3

SUMMARY:
The purpose of this study is to test different treatments to reduce relapse for drug-abusing adolescents who have completed family therapy. Adolescents receive 12 weeks of family therapy, designed to strengthen family relationships and develop skills for helping the adolescent avoid drug use. Then they are randomly assigned to receive one of three eight-week follow-up treatments: phone calls from a project therapist, group therapy, or a customized schedule of therapist visits with the adolescent, the adolescent's family and teachers, coaches, probation officers and others who can help the adolescent reach or maintain abstinence. Families are assessed using questionnaires and interviews before, during and after treatment, to provide information about family functioning, the adolescent's drug use, the adolescent's peers and other factors that may contribute to treatment success or failure. Adolescents also provide urine specimens for drug screening at assessment visits. Study investigators expect the study will show that a functional family environment and insulating adolescents from the influence of peers who use drugs will help prevent relapse for adolescents who have received family therapy.

ELIGIBILITY:
Inclusion Criteria:

1. At least one parent, step-parent, or surrogate parent willing to participate in the study
2. 13 to 18 years if age
3. meets DSM-IV (APA, 1994) diagnostic criteria for substance abuse or dependence
4. Lives in the Albuquerque metropolitan area or surrounding communities with a parent, step-parent, or surrogate parent; AND
5. Sufficient residential stability to permit probable contact at follow-up (e.g., not homeless at time of intake).

Exclusion Criteria:

1. Evidence of psychotic or organic state of sufficient severity to interfere with understanding of study instruments and procedures
2. Adolescent deemed dangerous to self or others during evaluation
3. Services other than outpatient treatment required for the adolescent (e.g., inpatient, detoxification)
4. Adolescent already has participated in treatment project at CFAR; AND
5. A sibling is already participating in project.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2004-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Drug use levels for adolescents who have received family therapy and one of the three aftercare regimens | pretx and 6 wks, 4 , 7 and 12 mos. post initial therapy session

CONTACTS AND LOCATIONS:
Overall Officials: Holly B. Waldron, Ph.D., Principal Investigator — Oregon Research Institute Center for Family and Adolescent Research (ORI/CFAR)
Locations (1):
- Oregon Res. Inst. Center for Family & Adolescent Research (CFAR), Albuquerque, New Mexico, United States